CLINICAL TRIAL: NCT04495569
Title: A Phase 1 Single Center, Parallel, Open Label Bridging Study to Evaluate on the Safety, Pharmacokinetic, Pharmacodynamics and Anti-drug Antibodies (ADA) of a Single Intramuscular Doses of SYN023 in Healthy Adult Subjects
Brief Title: A Bridging Study of the SYN023 on Healthy Adult Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synermore Biologics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYN023-005
Record Dates: First submitted 2020-05-10; First posted 2020-08-03 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2020-06

CONDITIONS: Communicable Disease Transmission; Zoonotic Disease; Rabies Human; Vaccine Reaction; Immunisation Reaction
Keywords: Bridging study; Rabies Vaccine; Monoclonal Antibody Cocktail; Biologics,
MeSH Terms: conditions — Zoonoses | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: Cohort A: Intramuscular 0.3 mg/kg SYN023 Cohort B: Intramuscular 0.3 mg/kg SYN023 + China licensed Vero Cell Rabies Vaccine (PEP)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group/Cohort A (Experimental): A single intramuscular injection of SYN023 at 0.3mg/kg
  Interventions: Biological: recombinant anti-rabies human monoclonal antibody injection (SYN023)
- Group/Cohort B (Experimental): A single intramuscular injection of SYN023 at 0.3mg/kg combined with the Chinese licensed Vero Cell Rabies Vaccine (following the PEP (Post-exposure Prophylaxis) recommendation)
  Interventions: Biological: recombinant anti-rabies human monoclonal antibody injection (SYN023); Biological: Rabies Vaccine

INTERVENTIONS:
Biological: recombinant anti-rabies human monoclonal antibody injection (SYN023) — The finished product of SYN023 is a mixture of two anti-rabies human monoclonal antibodies, CTB011 and CTB012 by equal quantity, containing 3.0 mg/mL active ingredients in both.
Biological: Rabies Vaccine — The Chinese licensed Vero Cell Freeze-dried Rabies Vaccine was injected to Cohort B as per the vaccination precedure on Days 1, 4, 8, 15, 28 respectively.
  Arms: Group/Cohort B

SUMMARY:
The Phase I bridging clinical trial is to evaluate on the safety, pharmacokinetics (PK), pharmacodynamics (PD) and ADA of a single intramuscular injection of recombinant anti-rabies human monoclonal antibody injection (SYN023) alone or combined with rabies vaccine in healthy subjects. The study primary purpose was to compare the pharmacokinetics (PK) between U.S and China subjects, therefore to lay a foundation for the follow-up clinical trials. The secondary purpose was to evaluate the PK, PD, Safety and ADA of SYN023 in Chinese Healthy subjects and compare with that of U.S. subjects.

DETAILED DESCRIPTION:
In this bridging study. the Pharmacodynamic, Pharmacokinetic, Safety and ADA(Anti-Drug Antibodies) were evaluated and compared between U.S. and China subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, fully understand the trial contents, process and possible adverse reactions, and cooperate to observe the adverse events;
2. Could participate the entire study according to the protocol;
3. Subjects including partners are willing to voluntarily take effective contraceptive measures from screening to 6 months after the last study drug administration.
4. Male and female healthy subjects aged 18-50 (including 18 and 50 years old)
5. The weight of male subjects shall not be less than 50 kg, and that of female subjects shall not be less than 45 kg and shall not be more than 90 kg. Body mass index (BMI) = body weight (kg) / height^2 (m^2), body mass index should be in the range of 18-30 kg/m2 (including);
6. Physical examination and vital signs are in normal range or the abnormality without clinical significance, and the body temperature is ≤ 37.6 °C.

Exclusion Criteria:

1. Smoked over 5 cigarettes per day for 3 months before the trial;
2. History of allergy (multi drugs and food allergy); history of severe allergic disease or allergic reaction; including allergy to any component of this drug;
3. History of alcohol addiction (14 units of alcohol per week: 1 unit = 285 mL beer, or 25 mL spirits, or 100 mL wine);
4. Blood donation or massive blood loss (> 450 mL) occurred within 3 months before screening;
5. History of autoimmune diseases;
6. History of chronic hepatitis ;
7. History of rabies virus infection;
8. Other acute or chronic diseases (within 6 months) that may interfere with the safety and efficacy evaluation of the subjects according to the investigator's judgment;
9. Receipt of an immunoglobulin or blood product within 90 days prior to study;
10. History of rabies vaccination;
11. Receipt of immunosuppressive medications included the inhaled or local immunosuppressant drugs within 45 days prior to Study;
12. Taken any prescribed, over-the-counter, vitamin product or herbal medicine within 14 days before screening;
13. Receipt of special diets (such as grapefruit) or endure strenuous physical exercise or any other factors affecting drug absorption, distribution, metabolism and excretion within 2 weeks before screening;
14. Had significant changes in diet or exercise habits recently;
15. Had been administrated with the investigational drug or participated in the clinical trial of the drug within three months before taking the investigational drug;
16. The evidence of clinically significant of the abnormalities of 12 lead ECG ;
17. Female subjects in lactation or positive for serum pregnancy test during screening for study;
18. Clinical significance of clinical laboratory results of screening, or suffered from the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardio cerebrovascular diseases within 6 months;
19. Positive in the screening of viral hepatitis (including hepatitis B and C), AIDS antibody, and treponema pallidum antibody;
20. Acute disease or drug administration from the screening to the initial of the study;
21. History of taken chocolate, or any food or drink containing caffeine or rich xanthine 24 hours prior to administration of the study drug;
22. History of taken any alcoholic product within 24 hours prior to administration of the study drug;
23. Drug abuse ;
24. Not suitable for enrolling in the study according to the investigator's judgment.

    Additional exclusion criteria for Group B:
25. Clinical significance of Immunoglobulin A abnormalities according to the investigator's judgment;
26. Undergoing anti-tuberculosis prophylaxis or treatment;
27. History of thyroidectomy, or treatment due to thyroid diseases in the past 12 months;
28. Diagnosed with serious angioneurotic edema in past 3 years or with the treatment in the past two years prior to the study;
29. Advanced tumors, or neoplasm in treatment and shows no evidence of recovery, or may relapse during the study;
30. No spleen or history of splenectomy;
31. Guillain-Barre syndrome or other serious neuropathy;
32. Receipt of live-attenuated vaccine within 30 days prior to the study;
33. Receipt of subunit or inactivated vaccine (such as pneumococcal vaccine), or allergy treatment within 14 days prior to the study;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
To compare the Tmax between Chinese and American subjects with a single dose of 0.3 mg/kg SYN023 alone or combined with rabies vaccine | 85 days
  Interval from time 0 to maximum measured concentration of CTB011 and CTB012 (SYN023 components) at Day1-0 h (pre-dose), Day1-6 h, Day2(24 h), Day3(48 h), Day4(72 h), Day6(120 h), Day8(168 h), Day15(336 h), Day29(672 h), Day36(840 h), Day43(1008 h), Day64(1512 h), Day85(2016 h) post-dose, using non compartmental analysis.
To compare the Cmax between Chinese and American subjects with a single dose of 0.3 mg/kg SYN023 alone or combined with rabies vaccine. | 85 days
  maximum concentration of CTB011 and CTB012 (SYN023 components) at Day1-0 h (pre-dose), Day1-6 h, Day2(24 h), Day3(48 h), Day4(72 h), Day6(120 h), Day8(168 h), Day15(336 h), Day29(672 h), Day36(840 h), Day43(1008 h), Day64(1512 h), Day85(2016 h) post-dose, using non compartmental analysis.
To compare the t1/2 between Chinese and American subjects with a single dose of 0.3 mg/kg SYN023 alone or combined with rabies vaccine. | 85 days
  The half life of CTB011 and CTB012 (SYN023 components) were estimated at Day1-0 h (pre-dose), Day1-6 h, Day2(24 h), Day3(48 h), Day4(72 h), Day6(120 h), Day8(168 h), Day15(336 h), Day29(672 h), Day36(840 h), Day43(1008 h), Day64(1512 h), Day85(2016 h) post-dose, using non compartmental analysis.
To compare the Clearance rate between Chinese and American subjects with a single dose of 0.3 mg/kg SYN023 alone or combined with rabies vaccine. | 85 days
  The clearance rate of CTB011 and CTB012 (SYN023 components) were estimated at at Day1-0 h (pre-dose), Day1-6 h, Day2(24 h), Day3(48 h), Day4(72 h), Day6(120 h), Day8(168 h), Day15(336 h), Day29(672 h), Day36(840 h), Day43(1008 h), Day64(1512 h), Day85(2016 h) post-dose, using non compartmental analysis.
SYN023 Monoclonal Antibody Areas Under the Curve (AUC0-last, AUC0-inf) for CTB011 and CTB012 | 85 days
  The area under the time concentration curve for SYN023 mAb components CTB011 and CTB012 were estimated at at Day1-0 h (pre-dose), Day1-6 h, Day2(24 h), Day3(48 h), Day4(72 h), Day6(120 h), Day8(168 h), Day15(336 h), Day29(672 h), Day36(840 h), Day43(1008 h), Day64(1512 h), Day85(2016 h) post-dose, using non compartmental analysis

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Event Incidence of healthy adult recipients of a single-dosed SYN023 0.3 mg/kg alone or combined with Rabies Vaccine | 85 days
  Electrocardiograms are performed to monitor subject safety. Laboratory evaluations for subject safety (adverse events) are serum chemistry evaluations, blood urea nitrogen, creatinine, bilirubin, alanine amino transferase, aspartate amino transferase, creatine phosphokinase, troponin, potassium, sodium, bicarbonate, calcium, complete blood count, platelet count, differential count, PT(prothrombin time, international normalized ratio) and PTT (partial prothrombin time and urinalyses for monitoring of safety. Additional laboratory tests may be required for evaluation of specific adverse events such as anaphylaxis and immune complex diseases. Adverse events were analyzed. A comparison of adverse event incidence between a single-dosed SYN023 0.3 mg/kg alone or combined with Rabies Vaccine were performed.
To evaluate the antibody protection level RVNA (Rabies Virus Neutralizing Antibodies)≥ 0.5 IU/mL of serum from healthy adult recipients of a single-dosed SYN023 0.3 mg/kg alone or combined with Rabies Vaccine | 85 days
  parallel the Cohort A and Cohort B to compare the antibody protection level (RVNA ≥ 0.5 IU/mL) between China and U.S. subjects
To evaluate the RVNA (Rabies Virus Neutralizing Antibodies) of serum from healthy adult recipients of a single-dosed SYN023 0.3 mg/kg alone or combined with Rabies Vaccine | 85 days
  parallel the Cohort A and Cohort B to compare the RVNA between China and U.S. subjects
To evaluate the ADA (Anti-Drug Antibodies) of serum from healthy adult recipients of a single-dosed SYN023 0.3 mg/kg alone or combined with Rabies Vaccine | 85 days
  parallel the Cohort A and Cohort B to compare the ADA between China and U.S. subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chao TY, Zhang SF, Chen L, Tsao E, Rupprecht CE. In Vivo Efficacy of SYN023, an Anti-Rabies Monoclonal Antibody Cocktail, in Post-Exposure Prophylaxis Animal Models. Trop Med Infect Dis. 2020 Feb 21;5(1):31. doi: 10.3390/tropicalmed5010031. PMID 32098049
- [Result] Chao TY, Ren S, Shen E, Moore S, Zhang SF, Chen L, Rupprecht CE, Tsao E. SYN023, a novel humanized monoclonal antibody cocktail, for post-exposure prophylaxis of rabies. PLoS Negl Trop Dis. 2017 Dec 20;11(12):e0006133. doi: 10.1371/journal.pntd.0006133. eCollection 2017 Dec. PMID 29261658
- [Result] Ding Y, Wu M, Zhang H, Zhu X, Hu Y, Li X, Liu J, Tsao E, Liu M, Li C. Safety, pharmacokinetics and pharmacodynamics of SYN023 alone or in combination with a rabies vaccine: An open, parallel, single dose, phase 1 bridging study in healthy Chinese subjects. Antiviral Res. 2020 Dec;184:104956. doi: 10.1016/j.antiviral.2020.104956. Epub 2020 Oct 19. PMID 33091433